CLINICAL TRIAL: NCT01384448
Title: A Randomized Trial Comparing Coronary CT Angiography and Stress Echocardiography for Evaluation of Low-to-Intermediate Risk Emergency Department Chest Pain Patients
Brief Title: Stress Echocardiography and Heart Computed Tomography (CT) Scan in Emergency Department Patients With Chest Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Jeffrey Levsky, Associate Director of Research, Department of Radiology, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MMC-11-03-107; 11SDG7380006 (Other Grant/Funding Number: American Heart Association National Center)
Record Dates: First submitted 2011-06-15; First posted 2011-06-29 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2017-03

CONDITIONS: Chest Pain; Angina; Angina Pectoris; Coronary Artery Disease
Keywords: stress echocardiography; coronary ct angiography
MeSH Terms: conditions — Chest Pain; Angina Pectoris; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Initial Stress Echocardiography (Experimental)
  Interventions: Procedure: Stress Echocardiography
- Initial Coronary CT Angiography (Experimental)
  Interventions: Procedure: Coronary CT Angiography

INTERVENTIONS:
Procedure: Stress Echocardiography — Stress echocardiography will be performed once. Treadmill stress is default. Patients that cannot exercise will receive dobutamine stress with or without atropine. Definity intravenous contrast will be given when needed.
  Other Names: stress echo; treadmill stress echocardiography; treadmill stress echo; exercise stress echocardiography; exercise stress echo; dobutamine stress echocardiography; dobutamine stress echo; ESE; TSE; DSE; SE
  Arms: Initial Stress Echocardiography
Procedure: Coronary CT Angiography — 64-detector, resting EKG-gated coronary CT angiography will be performed once. Patients with elevated heart rates will be given oral and/or intravenous metoprolol. Prospective gating with reduced tube current will be default. Retrospective gating with tube current modulation will be used in patients with higher heart rates.
  Other Names: Cardiac CT; Cardiac CTA; Coronary CT; Coronary CTA; Coronary Artery CT; Coronary Artery CTA; CT Angiography of the Coronary Arteries; Computed Tomography Angiography of the Coronary Arteries; CTA; CCT; CCTA
  Arms: Initial Coronary CT Angiography

SUMMARY:
The purpose of this study is to determine whether stress echocardiography or computed tomography (CT) of the heart is better at diagnosing emergency room chest pain patients to select appropriate candidates for hospitalization and further work-up.

ELIGIBILITY:
Inclusion Criteria:

* Presentation to the Emergency Department with chest pain
* Low-to-intermediate risk of coronary disease per Diamond-Forrester criteria
* Free of known coronary artery disease

Exclusion Criteria:

* Inability to undergo both stress echo or coronary CT for any reason
* Contraindication to intravenous iodinated contrast
* Dysrhythmia precluding EKG gating
* Heart rate greater than 60 with contraindication to beta blockers
* Administration of beta blockers within the last 12 hours
* Known severe cardiac valvular disease or pulmonary hypertension
* Stress echocardiography, coronary CT or catheterization within the last 6 months

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2011-08; Primary Completion 2016-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Hospital admission | 30 days

SECONDARY OUTCOMES:
Emergency Department length of stay | 30 days
Hospital length of stay | 30 days
Estimated cost of initial care | 30 days
Repeat visits to the Emergency Department | 30 days and 1 year
Death | 30 days and 1 year
Non-fatal myocardial infarction | 30 days and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M Levsky, MD, PhD, Principal Investigator — Montefiore Medical Center/Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center - Weiler / Einstein Division, The Bronx, New York, United States

REFERENCES:
- [Background] Levsky JM, Haramati LB, Taub CC, Spevack DM, Menegus MA, Travin MI, Vega S, Lerer R, Brown-Manhertz D, Hirschhorn E, Tobin JN, Garcia MJ. Rationale and design of a randomized trial comparing initial stress echocardiography versus coronary CT angiography in low-to-intermediate risk emergency department patients with chest pain. Echocardiography. 2014 Jul;31(6):744-50. doi: 10.1111/echo.12464. Epub 2013 Dec 23. PMID 24372760
- [Background] Levsky JM, Haramati LB, Spevack DM, Menegus MA, Chen T, Mizrachi S, Brown-Manhertz D, Selesny S, Lerer R, White DJ, Tobin JN, Taub CC, Garcia MJ. Coronary Computed Tomography Angiography Versus Stress Echocardiography in Acute Chest Pain: A Randomized Controlled Trial. JACC Cardiovasc Imaging. 2018 Sep;11(9):1288-1297. doi: 10.1016/j.jcmg.2018.03.024. Epub 2018 Jun 13. PMID 29909113